CLINICAL TRIAL: NCT00900874
Title: Comparing Rapid Bronchodilatory Effect of Formoterol and Salbutamol in Children Between 5-15 Years With Mild to Moderate Acute Exacerbation of Asthma- A Double Blind Randomized Controlled Trial
Brief Title: Rapid Onset Action of Salbutamol Versus Formoterol
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: J.Jenish Rajma, AIIMS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIIIMS
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2009-05-13 (Estimated); Status verified 2009-05

CONDITIONS: Bronchial Asthma
Keywords: Formoterol; Rapid bronchodilation
MeSH Terms: conditions — Asthma | interventions — Albuterol; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Salbutamol + steroid
  Interventions: Drug: salbutamol
- 2 (Active Comparator): Formoterol + steroid
  Interventions: Drug: Formoterol

INTERVENTIONS:
Drug: salbutamol — two puffs (100 microgram each of salbutamol) by MDI and spacer
  Arms: 1
Drug: Formoterol — Formoterol 2 puffs (6 µg /puff) by MDI and spacer
  Arms: 2

SUMMARY:
The hypothesis of this study is that the onset of rapid bronchodilatory effect of inhaled Formoterol (12 microgram) is comparable to that of inhaled salbutamol (200 microgram) i.e., the difference in mean forced expiratory volume in 1 second (FEV1) between the 2 groups at 1, 5, 10, 30 and 60 minutes will be less than 10% in children between 5-15 years with mild acute exacerbation of asthma.

DETAILED DESCRIPTION:
It is desirable to have a single MDI that can be used as both LABA and SABA. There are few studies involving few children on use of formoterol that shows rapid bronchodilatation in children with asthma and no study that used it as rescue drug in children with acute exacerbation of asthma. The purpose of the present study is to evaluate whether the rapid bronchodilatory effect of formoterol is similar to that of salbutamol in children of 5-15 years with mild exacerbation of asthma.

Children will receive either salbutamol or formoterol by MDI. Participants will be explained about the study, spirometry and inhalation of medicine with MDI and spacer. Children will receive two puffs (100 microgram each of salbutamol) or Formoterol 2 puffs (6µg /puff) by MDI and spacer. Each child will be explained about the inhalation technique by using a MDI of placebo. After shaking the MDI it will be attached to spacer (700ml volume) and actuated. Child will be asked to take 5 tidal breaths. Another puff will be given by similar method.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 5-15 years of either sex seeking treatment with mild exacerbation of asthma in pediatric chest clinic or Pediatric OPD
2. Mild exacerbation will be defined as:

   * children presenting with increase in symptoms (cough, wheeze, breathlessness) for less than 7 days duration
   * no chest indrawing
   * no difficulty in speech
   * clinical asthma score (or pulmonary index score-annexure 1) between 6-9

Exclusion Criteria:

1. Children with life threatening asthma detected by presence of any of the following:

   * severe chest indrawing
   * cyanosis
   * irregular respiration
   * altered sensorium
2. Children with other chronic respiratory conditions like tuberculosis, cystic fibrosis or other acute illness that would complicate current treatment and response for asthma
3. If child has taken salbutamol in last 6 hours or if he is on long acting beta agonists (formoterol or salmeterol)
4. Child not able to perform spirometry
5. Parents refusing to give consent

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Difference in mean FEV1 between the two groups at 1, 5, 10, 30, 60 minutes | 60 min

SECONDARY OUTCOMES:
Difference in average clinical asthma score between two groups | 60 min
Adverse effects like tremors, vomiting, palpitation, etc, in two groups | 60 mins
Number of patients requiring hospitalization in two groups at end of study period in two groups | 60 min

CONTACTS AND LOCATIONS:
Locations (1):
- AIIMS, New Delhi, New Delhi, India

REFERENCES:
- [Derived] Arun JJ, Lodha R, Kabra SK. Bronchodilatory effect of inhaled budesonide/formoterol and budesonide/salbutamol in acute asthma: a double-blind, randomized controlled trial. BMC Pediatr. 2012 Mar 7;12:21. doi: 10.1186/1471-2431-12-21. PMID 22394648